CLINICAL TRIAL: NCT00409825
Title: A Study of the Pharmacology of 17-Hydroxyprogesterone Caproate in Pregnancy
Brief Title: Study of Pharmacology of 17-OHPC in Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #0603056; 5U10HD047905-02 (NIH)
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy
MeSH Terms: interventions — 17-alpha-Hydroxyprogesterone; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Part 1 (Experimental): Part 1 done after 4 weekly 17-OHPC injections completed, between 20 6/7 to 24 6/7 weeks gestation. 10 cc blood drawn pre-5th injection. 10 cc blood drawn 12 hours post-dose and 7 consecutive days. 24-hour urine collected days 4-5 within 7 days post-injection. Part 2 done 31 0/7 to 34 6/7 or at 35 0/7 weeks. 10 cc blood drawn pre weekly injection, 12 hours post-dose, and 7 consecutive days. 24-hour urine collected between days 4-5 within 7 days post-injection. A subject in whom Part 2 is performed during the last scheduled injection of 17-OHPC (at or around 35 0/7 weeks) will have the option to participate in Part 3, in which 10 cc of blood will be drawn serially over 21 days after completing Part 2. Blood will be drawn on days 9, 11, 14, 17, 20, 24, 28 after the last injection. Part 4: At the time of labor and delivery, subject will have 10cc of blood removed from a maternal peripheral vein. 10cc of blood will be collected from the placenta/umbilical cord after delivery.
  Interventions: Drug: 17-OHPC; Procedure: Blood Draws

INTERVENTIONS:
Drug: 17-OHPC — Intra-muscular injection of 250 mg 17-OHPC administered weekly between the second and third trimesters of pregnancy, until time of delivery.
  Other Names: 17-alpha-hydroxyprogesterone caproate
Procedure: Blood Draws — 10 cc of blood will be drawn prior to the fifth weekly administration of 17-OHPC during second trimester of pregnancy, and then once daily for seven consecutive days post-dose. 10 cc of blood also will be drawn prior to weekly administration of 17-OHPC from sixth weekly dose in the second trimester until the last scheduled dose in the third trimester. Prior to this last scheduled dose, 10 cc of blood will be drawn, as well as once daily for seven consecutive days post-dose.

SUMMARY:
We are examining the pharmacology of 17-OHPC in pregnancy, specifically between the second and third trimesters.

DETAILED DESCRIPTION:
The recently completed trial by the National Institute of Child Health and Human Development (NICHD)-sponsored Maternal-Fetal Medicine Units (MFMU) Network has demonstrated that intramuscular 17-alpha-hydroxyprogesterone caproate (17-OHPC) substantially reduces the rate of preterm birth in women at high risk for preterm delivery because of a prior spontaneous preterm birth. No other strategy or treatment for prevention of preterm birth has proven to be effective. Consequently, the American College of Obstetricians and Gynecologists has cautiously supported this treatment but points out that much more information about this therapy and alternative therapies is required. Although a large body of evidence exists about the safety of this treatment, almost nothing is known about the pharmacology of this agent, especially in pregnancy. The purpose of this study is to define the pharmacology of 17-hydroxyprogesterone caproate in pregnancy. This protocol will focus on pharmacokinetics and placental transport and provide preliminary data on the pharmacoepidemiology of 17-OHPC. The primary research question of this study is: Do the pharmacokinetics of 17-OHPC as represented by area under the concentration vs. time curve after IM injection of 250 mg 17-OHPC differ between the second and third trimesters of pregnancy? We will obtain blood samples prior to and daily for one week after injection of 17-OHPC (8 samples total) for each of two parts of the study, with an optional third part for eligible subjects. Additionally, blood samples will be collected prior to each weekly injection of the study drug and at time of delivery. Approximately 60 subjects (ages 18-45) will be accrued at one of the Obstetrical Fetal Pharmacology Research Units (OPRU) Network sites, with 15 at Magee-Womens Hospital of the University of Pittsburgh Medical Center. Study treatment will be administered until delivery. The total duration of this multi-center study is 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation prior to 20 0/7 weeks gestation
* Planning to receive or receiving 17-OHPC (250 mg IM weekly)
* Previous history of preterm birth
* Able to give consent

Exclusion Criteria:

* Fetal demise, anomaly, or growth restriction
* Hepatic or renal dysfunction
* Placental previa or abruptio placenta
* Polyhydramnios/oligohydramnios
* Short cervix or planned cerclage
* Chronic use of steroids, antiepileptics, antihypertensives, SSRS, street drugs
* Participation in another interventional study that influences gestational age at delivery
* Heparin treatment of known platelet count <100,000/mm3 (because of contraindication to intra-muscular injections)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve N. Caritis, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Georgetown University, Washington D.C., District of Columbia
  - Magee-Womens Hospital of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas, Galveston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] ACOG News Release: Progesterone recommended in certain high risk pregnancies to help prevent preterm birth. October 31, 2003
- [Background] Onsrud M, Paus E, Haug E, Kjorstad K. Intramuscular administration of hydroxyprogesterone caproate in patients with endometrial carcinoma. Pharmacokinetics and effects on adrenal function. Acta Obstet Gynecol Scand. 1985;64(6):519-23. doi: 10.3109/00016348509156732. PMID 2932883
- [Background] Kiesling H, Elmquist A: Acta Endocrinol 28:502, 1958
- [Background] GASSNER FX, MARTIN RP, SHIMODA W, ALGEO JW. Metaolism of radioactive steroid esters in the bovine male and female. Fertil Steril. 1960 Jan-Feb;11:49-73. doi: 10.1016/s0015-0282(16)33663-9. No abstract available. PMID 13826776
- [Background] LANGECKER H, HARWART A, JUNKMANN K. [1-Phenyl-propanol as a choleretic]. Naunyn Schmiedebergs Arch Exp Pathol Pharmakol. 1955;225(4):303-8. No abstract available. German. PMID 13253659
- [Background] WIENER M, LUPU CI, PLOTZ EJ. Metabolism of 17 alpha-hydroxyprogesterone-4-C14-17 alpha-caproate by homogenates of rat liver and human placenta. Acta Endocrinol (Copenh). 1961 Apr;36:511-9. No abstract available. PMID 13785108
- [Background] Endocrinology & human gestation. IN: Reproductive Endocrinology, p458. Edited by EY Adashi, Lippincott-Raven Publishers, Philadelphia, PA 1996.
- [Background] Challis JRG, Matthews SG, Gibb W, Lye SJ. Endocrine and paracrine regulation of birth at term and preterm. Endocr Rev. 2000 Oct;21(5):514-50. doi: 10.1210/edrv.21.5.0407. PMID 11041447
- [Background] Johnson JW, Lee PA, Zachary AS, Calhoun S, Migeon CJ. High-risk prematurity--progestin treatment and steroid studies. Obstet Gynecol. 1979 Oct;54(4):412-8. PMID 492618
- [Background] Keirse MJ. Progestogen administration in pregnancy may prevent preterm delivery. Br J Obstet Gynaecol. 1990 Feb;97(2):149-54. doi: 10.1111/j.1471-0528.1990.tb01740.x. PMID 2138496
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Background] Csapo AI. The 'see-saw' theory of parturition. Ciba Found Symp. 1977;(47):159-210. No abstract available. PMID 246391
- [Background] Haluska GJ, Wells TR, Hirst JJ, Brenner RM, Sadowsky DW, Novy MJ. Progesterone receptor localization and isoforms in myometrium, decidua, and fetal membranes from rhesus macaques: evidence for functional progesterone withdrawal at parturition. J Soc Gynecol Investig. 2002 May-Jun;9(3):125-36. PMID 12009386
- [Background] Lye S: Personal communication
- [Background] JUNKMANN K. [Estrogens with prolonged action]. Naunyn Schmiedebergs Arch Exp Pathol Pharmakol. 1953;220(5):358-64. No abstract available. Undetermined Language. PMID 13144797
- [Background] KESSLER WB, BORMAN A. Some biological activities of certain progestogens. I. 17 alpha-Hydroxyprogesterone 17-n-caproate. Ann N Y Acad Sci. 1958 Jul 30;71(5):486-93. doi: 10.1111/j.1749-6632.1958.tb46779.x. No abstract available. PMID 13583805
- [Background] JOHNSTONE EE, FRANKLIN RR. ASSAY OF PROGESTINS FOR FETAL VIRILIZING PROPERTIES USING THE MOUSE. Obstet Gynecol. 1964 Mar;23:359-62. No abstract available. PMID 14128463
- [Background] SUCHOWSKY G, JUNKMANN K. [Research on the maintenance of pregnancy by 17 alpha-hydroxyprogesterone caproate in the castrated pregnant rabbit]. Acta Endocrinol (Copenh). 1958 Jun;28(2):129-31. No abstract available. German. PMID 13532385
- [Background] Courtney KD, Valerio DA. Teratology in the Macaca mulatta. Teratology. 1968 May;1(2):163-72. doi: 10.1002/tera.1420010205. No abstract available. PMID 4321743
- [Background] Carbone JP, Brent RL. Genital and nongenital teratogenesis of prenatal progestogen therapy: the effects of 17 alpha-hydroxyprogesterone caproate on embryonic and fetal development and endochondral ossification in the C57B1/6J mouse. Am J Obstet Gynecol. 1993 Nov;169(5):1292-8. doi: 10.1016/0002-9378(93)90296-u. PMID 8238197
- [Background] Seegmiller RE, Nelson GW, Johnson CK. Evaluation of the teratogenic potential of delalutin (17 alpha-hydroxyprogesterone caproate) in mice. Teratology. 1983 Oct;28(2):201-8. doi: 10.1002/tera.1420280208. PMID 6648824
- [Background] Varma TR, Morsman J. Evaluation of the use of Proluton-Depot (hydroxyprogesterone hexanoate) in early pregnancy. Int J Gynaecol Obstet. 1982 Feb;20(1):13-7. doi: 10.1016/0020-7292(82)90039-x. PMID 6126401
- [Background] Michaelis J, Michaelis H, Gluck E, Koller S. Prospective study of suspected associations between certain drugs administered during early pregnancy and congenital malformations. Teratology. 1983 Feb;27(1):57-64. doi: 10.1002/tera.1420270109. PMID 6845218
- [Background] Resseguie LJ, Hick JF, Bruen JA, Noller KL, O'Fallon WM, Kurland LT. Congenital malformations among offspring exposed in utero to progestins, Olmsted County, Minnesota, 1936-1974. Fertil Steril. 1985 Apr;43(4):514-9. doi: 10.1016/s0015-0282(16)48490-6. PMID 3987922
- [Background] Check JH, Rankin A, Teichman M. The risk of fetal anomalies as a result of progesterone therapy during pregnancy. Fertil Steril. 1986 Apr;45(4):575-7. doi: 10.1016/s0015-0282(16)49292-7. PMID 3956772
- [Background] Katz Z, Lancet M, Skornik J, Chemke J, Mogilner BM, Klinberg M. Teratogenicity of progestogens given during the first trimester of pregnancy. Obstet Gynecol. 1985 Jun;65(6):775-80. PMID 3158848
- [Background] Kester PA. Effects of prenatally administered 17 alpha-hydroxyprogesterone caproate on adolescent males. Arch Sex Behav. 1984 Oct;13(5):441-55. doi: 10.1007/BF01541429. PMID 6517685
- [Background] Schardein JL. Congenital abnormalities and hormones during pregnancy: a clinical review. Teratology. 1980 Dec;22(3):251-70. doi: 10.1002/tera.1420220302. PMID 7015547
- [Background] Raman-Wilms L, Tseng AL, Wighardt S, Einarson TR, Koren G. Fetal genital effects of first-trimester sex hormone exposure: a meta-analysis. Obstet Gynecol. 1995 Jan;85(1):141-9. doi: 10.1016/0029-7844(94)00341-a. PMID 7800312
- [Background] Reprotox Database. Hydroxyprogesterone 17-. Reprotox. org. March 1, 2003.
- [Background] Florey K: Hydroxyprogesterone caproate. IN: Analytical profiles of drug substances. Vol 4. 208-224 Editors: Academic Press, NY, NY, 1975.
- [Background] REIFENSTEIN EC Jr. Introduction of marked as well as prolonged biologic activity by esterification; 17-alpha-hydroxyprogesterone caproate, a unique progestational compound. Fertil Steril. 1957 Jan-Feb;8(1):50-79. doi: 10.1016/s0015-0282(16)32585-7. No abstract available. PMID 13405048
- [Background] Karalis K, Goodwin G, Majzoub JA. Cortisol blockade of progesterone: a possible molecular mechanism involved in the initiation of human labor. Nat Med. 1996 May;2(5):556-60. doi: 10.1038/nm0596-556. PMID 8616715
- [Background] Hvilsom GB, Thorsen P, Jeune B, Bakketeig LS. C-reactive protein: a serological marker for preterm delivery? Acta Obstet Gynecol Scand. 2002 May;81(5):424-9. doi: 10.1034/j.1600-0412.2002.810509.x. PMID 12027816
- [Background] Mackler AM, Iezza G, Akin MR, McMillan P, Yellon SM. Macrophage trafficking in the uterus and cervix precedes parturition in the mouse. Biol Reprod. 1999 Oct;61(4):879-83. doi: 10.1095/biolreprod61.4.879. PMID 10491619

RESULTS

PARTICIPANT FLOW:
Groups:
- AUC1 vs AUC2: AUC 1 done after 4 weekly 17-OHPC injections completed, between 20 6/7 to 24 6/7 weeks gestation. 10 cc blood drawn pre-5th injection. 10 cc blood drawn 12 hours post-dose and 7 consecutive days. 24-hour urine collected days 4-5 within 7 days post-injection.
  AUC 2 done 31 0/7 to 34 6/7 or at 35 0/7 weeks. 10 cc blood drawn pre weekly injection, 12 hours post-dose, and 7 consecutive days. 24-hour urine collected between days 4-5 within 7 days post-injection.
Period: Overall Study
Arm/Group | AUC1 vs AUC2
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AUC1 vs AUC2
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.01 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 18
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in the Area Under the Concentration vs. Time Curve in the Second and Third Trimesters of Pregnancy.
Description: Change in the area under the concentration vs. time curve in the second and third trimesters of pregnancy.
  We compared AUC at each PK study visit. Measurements were obtained at 0, 1, 2, 3, 4, 5, 6, 7 days.
Time Frame: Second and third trimesters of pregnancy
Measure: Mean (Standard Deviation); unit: ng/ML/day
Groups:
- Part 1: Part 1 done after 4 weekly 17-OHPC injections completed, between 20 6/7 to 24 6/7 weeks gestation. 10 cc blood drawn pre-5th injection. 10 cc blood drawn 12 hours post-dose and 7 consecutive days. 24-hour urine collected days 4-5 within 7 days post-injection. Part 2 done 31 0/7 to 34 6/7 or at 35 0/7 weeks. 10 cc blood drawn pre weekly injection, 12 hours post-dose, and 7 consecutive days. 24-hour urine collected between days 4-5 within 7 days post-injection.
Arm/Group | Part 1
Number analyzed (Participants) | 61
ng/ML/day
  AUC -1 | 115 (44)
  AUC - 2 | 136 (52)

ADVERSE EVENTS:
Groups:
- Part 1: Part 1 done after 4 weekly 17-OHPC injections completed, between 20 6/7 to 24 6/7 weeks gestation. 10 cc blood drawn pre-5th injection. 10 cc blood drawn 12 hours post-dose and 7 consecutive days. 24-hour urine collected days 4-5 within 7 days post-injection. Part 2 done 31 0/7 to 34 6/7 or at 35 0/7 weeks. 10 cc blood drawn pre weekly injection, 12 hours post-dose, and 7 consecutive days. 24-hour urine collected between days 4-5 within 7 days post-injection. A subject in whom Part 2 is performed during the last scheduled injection of 17-OHPC (at or around 35 0/7 weeks) will have the option to participate in Part 4, in which 10 cc of blood will be drawn serially over 21 days after completing Part 2. Blood will be drawn on days 9, 11, 14, 17, 20, 24, 28 after the last injection. Part 3: At the time of labor and delivery, subject will have 10cc of blood removed from a maternal peripheral vein. 10cc of blood will be collected from the placenta/umbilical cord after delivery.
Arm/Group | Part 1
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No